CLINICAL TRIAL: NCT02559882
Title: Testing Effectiveness of Renal Denervation in Patients With Therapy-resistant Hypertension
Brief Title: How to Test Success of a Renal Denervation
Status: Terminated | Type: Observational
Why Stopped: The Enterprise decided to stop the production of the catheter used for the clinical indicated renal denervation
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: EK2015_0045
Record Dates: First submitted 2015-08-24; First posted 2015-09-25 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Hypertension, Resistant to Conventional Therapy
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study aimed to assess the success of a clinically indicated renal denervation by different tests and correlate the results of the tests with the clinical outcome.

DETAILED DESCRIPTION:
We aim to test the response to adenosine infusion, cold pressure test, flow mediated dilation of renal artery before and after a clinical indicated renal denervation. Renal Denervation is not a study intervention

ELIGIBILITY:
Inclusion Criteria:

Male and female patients 18 years to 85 years of age, with a diagnosis of re-sistant hypertension (office sitting blood pressure >140/90 mmHg and 24-hour blood pressure >130/80 mmHg in patients treated with at least three antihypertensive drugs including a diuretic) and a clinical indication for a renal denervation.

Exclusion Criteria:

* Secondary cause of hypertension
* Anatomical contraindication to renal denervation (renal artery diameter less than 4 mm or more than 8 mm), multiple renal artery, length to bifurcation less than 2 cm
* Heart failure (normal ejection fractions on echocardiography and no clinical signs and symptoms of heart failure).
* Alcohol or drug abuse,
* Malignancy (unless healed or remission > 5 years)
* Pregnancy
* Know allergy to contrast medium
* Participation in another study within the last month

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with therapy resistant hypertension and clinical indication for renal nerve ablation
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2015-08; Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Response to adenosine infusion, cold pressure test, flow mediated dilation of renal artery before and 1 year after renal denervation B | chronic
  Changes in blood pressure and heart rate, in renal artery diameter and flow during adenosine infusion before and 1 year after renal denervation
lood pressure (office and 24-hour blood pressure), laboratory parameter before and 12 months after catheter-based renal denrevation | chronic

SECONDARY OUTCOMES:
Blood pressure (office and 24-hour blood pressure), laboratory parameter before and 1, 3, 6 months after catheter-based | chronic
  Blood pressure (office and 24-hour blood pressure), laboratory parameter before and 1, 3, 6 months after catheter-based

CONTACTS AND LOCATIONS:
Overall Officials: Isabella Sudano, MD Phd, Principal Investigator — University Heart Center Cardiology University Hospital Zurich
Locations (1):
- Department of Cardiology University Heart Center Zurich University Hospital, Zurich, Switzerland